CLINICAL TRIAL: NCT03106337
Title: A Multivariate Analysis of Factors Predictive of Carcinoma in Follicular Neoplasms of the Thyroid Gland
Brief Title: Diagnostic Accuracy of Shear-Wave Elastography for the Preoperative Risk Stratification of Follicular Lesions of the Thyroid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Antonia Stephen, MD, Assistant Professor of Surgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007P001161
Record Dates: First submitted 2014-04-25; First posted 2017-04-10 (Actual); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Thyroid Nodule; Follicular Neoplasm
Keywords: Thyroid; Follicular Neoplasms; Bethesda System; Elastography; Doppler ultrasound; Thyroidectomy
MeSH Terms: conditions — Thyroid Nodule; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Shear-Wave Elastography (Experimental): Shear-Wave Elastography was performed on patients scheduled for partial/total thyroidectomy. Results were compared with pathology from surgical excision.
  Interventions: Device: Shear-Wave Elastography

INTERVENTIONS:
Device: Shear-Wave Elastography — Shear-Wave Elastography was performed on patients scheduled for partial/total thyroidectomy. Results were compared with pathology from surgical excision.
  Other Names: Supersonic Aixplorer

SUMMARY:
As many as 70-85% subjects diagnosed with a follicular lesion on biopsy and undergoing surgery will have benign lesions verified by histopathology after surgery.

Currently there is no method of pre-operatively diagnosing benign follicular lesions, as a result these subjects will have had surgery for diagnosis of a benign lesion.

The aim of this study is to see whether shear-wave elastography, a new ultrasound technology can help pre-operatively diagnose benign follicular lesions. If successful, a lot of patients will not need surgery for the diagnosis of a benign lesion.

The main goal of this study will be to evaluate the diagnostic accuracy of a new ultrasound technology, shear-wave elastography (SWE), for the diagnosis of malignancy in follicular lesions. Participants who have been diagnosed with a follicular lesion on thyroid biopsy and are scheduled for thyroid surgery will be eligible to participate. All participants will undergo a detailed ultrasound examination prior to their surgery. The results of the ultrasound will be compared with histopathology after surgery to test the diagnostic accuracy of SWE.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a Follicular Neoplasm on fine needle aspiration biopsy
* Patients >18 years of age

Exclusion Criteria

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonia E. Stephen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Samir AE, Dhyani M, Anvari A, Prescott J, Halpern EF, Faquin WC, Stephen A. Shear-Wave Elastography for the Preoperative Risk Stratification of Follicular-patterned Lesions of the Thyroid: Diagnostic Accuracy and Optimal Measurement Plane. Radiology. 2015 Nov;277(2):565-73. doi: 10.1148/radiol.2015141627. Epub 2015 May 7. PMID 25955578

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shear-Wave Elastography
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Shear-Wave Elastography
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Shear-Wave Elastography (SWE) Values in kiloPascals (kPa)
Description: Elastography provides a quantitative score of thyroid nodule stiffness that is expected to correlate with the biological nature of the nodule. Mean SWE values, in three planes: traverse plane, sagittal plane and transverse plane with nodule in the center, of all benign lesions were compared with mean SWE values of all malignant lesions on histopathology obtained post surgery.
Time Frame: Baseline (Day 0)
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: kPa
Groups:
- Shear-Wave Elastography, Benign Lesions: Shear-Wave Elastography was performed on patients scheduled for partial/total thyroidectomy. Results were compared with pathology from surgical excision. This cohort includes all participants with benign lesions.
- Shear-Wave Elastography, Malignant Lesions: Shear-Wave Elastography was performed on patients scheduled for partial/total thyroidectomy. Results were compared with pathology from surgical excision. This cohort Includes all participants with malignant lesions.
Arm/Group | Shear-Wave Elastography, Benign Lesions | Shear-Wave Elastography, Malignant Lesions
Number analyzed (Participants) | 24 | 11
kPa
  Transverse Plane | 17.50 (7.65) | 31.03 (13.54)
  Sagittal Plane | 23.64 (14.86) | 32.14 (11.98)
  Transverse Plane with Nodule in the Center | 17.89 (9.1) | 33.80 (12.50)

ADVERSE EVENTS:
Arm/Group | Shear-Wave Elastography
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes